CLINICAL TRIAL: NCT07025083
Title: Adaptation of Family Check-Up Online in the Latinx Community to Reduce Youth Substance Use
Brief Title: Adaptation of the Family Check-Up Online
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 33365; 1R34DA061150-01 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-06-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-04

CONDITIONS: Substance Use (Drugs, Alcohol)
Keywords: adolescence; parenting; adaptation; family; substance use intent
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family Check-Up Online Adapted for Latinx Families (Experimental): In this arm, participants will receive the Family Check-Up Online adapted for Latinx families plus telehealth support from a promotore de salud.
  Interventions: Behavioral: Adapted Family Check-Up Online
- Original Family Check-Up Online (Experimental): In this arm, participants will receive the original Family Check-Up online in Spanish.
  Interventions: Behavioral: Original Family Check-Up Online
- Waitlist Control (No Intervention): The waitlist control group will not receive the intervention during the trial, but will have the option to participate in the Family Check-Up Online after the trial is over.

INTERVENTIONS:
Behavioral: Adapted Family Check-Up Online — The Family Check-Up Online is a digital intervention that includes an assessment, computer-generated feedback, and intervention modules that focus on improving family relationships and parenting skills in order to reduce child mental health problems and to improve child self-regulation. These modules include Healthy Behaviors for Stressful Times, Positive Parenting, Rules and Consequences, Supporting School Success, and Communication. In addition, two modules for Latinx families are being added in the adapted version. This version represents a deep adaptation.
  Arms: Family Check-Up Online Adapted for Latinx Families
Behavioral: Original Family Check-Up Online — This version is the original Family Check Up Online translated into Spanish without the adaptions. This represents a surface-level adaptation.
  Arms: Original Family Check-Up Online

SUMMARY:
Latinx people are the largest and fastest growing minority population in the U.S., yet most lack access to community responsive preventative interventions to reduce substance use among youth. Effective implementation of evidence-based interventions that can be delivered online is critical to reduce substance use and problem behaviors among ethnic populations and to scale up for broad dissemination. Adaptation to address community needs has improved parenting practices and youth outcomes beyond the original evidence-based parenting interventions, and adapted parenting programs have the potential to improve cultural socialization, which is associated with improved behavioral outcomes among Latinx youth. However, ongoing tensions in the field highlight the question of whether deep adaptations compared to surface-level adaptations (e.g., translation only) are needed. The FCU is an evidence-based parenting program that has a strong history of reducing substance abuse and externalizing symptoms (e.g., problem behaviors). A community-based participatory approach will be employed to culturally adapt the FCU Online and identify implementation strategies to improve access to and adoption of the intervention, leveraging community and resiliency-promoting assets. Promotores de salud, Spanish-speaking community health workers in an existing community-based research network will deliver the program. To reach the goals of the study, the following aims will guide this research. In Aim 1, a community advisory board of 6 parents and 6 promotores de salud will meet monthly to guide the ecological adaptation of the FCU Online modules and implementation strategies with promotores. In Aim 2, the online version of the intervention will be adapted using iterative Plan-Do-Study-Act cycles to get usability feedback from members of the community advisory board, consistent with best practices designed to adapt interventions in community settings. In Aim 3, using a Hybrid 1, mixed methods design, researchers will assess feasibility, accessibility, adoption, and potential effectiveness of the adapted intervention, FCU-L Online. The team will recruit 108 Latinx families into a 3-arm wait-list randomized control trial: n=36 in the culturally adapted FCU-L Online (e.g., deep adaptation), n=36 in the FCU Online in Spanish without adaptation (e.g., surface level adaptation), and n= 36 in a waitlist control group. Feasibility, accessibility, and adoption will be assessed according to quantitative benchmarks, and qualitative feedback will assess the barriers and facilitators of implementation. Potential effectiveness will be assessed (p < .15), including improvement of key intervention mechanisms (parenting practices, parenting efficacy, and cultural socialization) as well as child outcomes (substance use, intentions to use, and externalizing behavior). Findings from this study will inform a Hybrid II randomized controlled implementation trial to test effectiveness while scaling up dissemination of the FCU-L Online. This research could ultimately reduce lifetime risk for substance use among Latinx youth by improving parenting practices and supporting cultural socialization.

DETAILED DESCRIPTION:
In this study the investigators propose the following specific aims:

1. Employ community perspectives to adapt and maximize feasibility, acceptability, and adoption of the online Spanish-speaking version of Family Check-Up among Latinx families. A group of 12 parents of middle school youth (n=6) and stakeholders, including promotores (n=6), will meet monthly in the first year to guide user-informed adaptations that incorporate Latinx community perspectives into the content and delivery processes.
2. Develop a adapted version of Family Check-Up Online for Latinx families (FCU-L Online). Adapt current modules and develop two community responsive modules to address key issues identified by parents and stakeholders. Iterative usability feedback with an additional set of Spanish-speaking parents and stakeholders (N=12) will inform development in two Plan-Do-Study-Act (PDSA) cycles, consistent with best practices designed to adapt interventions in community settings. Additionally, adaptations to the implementation process using PDSA cycles will be made to support delivery by promotores.
3. Conduct a Hybrid 1 pilot study to evaluate the feasibility, acceptability, adoption, and potential effectiveness of FCU-L Online delivered by promotores, focusing on parenting practices as the mechanism of action. We will randomize 108 Spanish-speaking Latinx families with a youth aged 11-14 years to the adapted intervention delivered by promotores, the Spanish FCU Online without adaptation delivered by the research team, or a wait-list control.

Goal 1: Assess feasibility, acceptability, and adoption of the adapted FCU Online with new content (e.g., how the past affects parenting, developing cultural strength) and implementation strategies: surveys (N=108; e.g., acceptability, socialization) and interviews with a subset of parents (N=6) and promotores (N=6).

Goal 2: Evaluate the potential effectiveness of the adapted FCU Online on the primary outcomes, parenting practices (e.g., parenting efficacy, positive parenting, socialization) and explore effects on youth outcomes (e.g., substance use/intent and externalizing behavior).

ELIGIBILITY:
Parent Inclusion Criteria:

* being a self-identified Latinx parent or guardian of a youth age 11-14
* speaking Spanish
* cognitively able to complete a brief screener
* assessments at a 6th grade reading level
* willing to participate in an online intervention
* willing for their child to complete confidential assessments

Youth Inclusion Criteria:

* being a middle school student age 11-14
* reading at the 2nd grade level in English or Spanish

Exclusion Criteria:

* having low concerns on the Positive Family Support screener

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Telehealth Usability Questionnaire | 3 months
  We will use the Telehealth Usability Questionnaire(TUQ) to assess the quality of the program's technology interface and telehealth interaction. TUQ includes 21 items and covers five domains of telehealth system usability: usefulness (3 items; e.g., "FCU Online improves my access to health and preventative services"), ease of use and learnability (3 items; e.g., "It was simple to use this system"), interface quality (4 items; e.g., "The way I interact with this system is pleasant"), interaction quality (4 items; e.g., "I could easily talk to the coach using the telehealth system"), reliability (3 items; e.g., "Whenever I made a mistake using the system, I could recover easily and quickly"), and satisfaction and future use (4 items; e.g., "I feel comfortable communicating with the coach using the telehealth system"). All TUQ subscales have shown good internal consistency (Cronbach's αs > 0.8) and have been validated in Spanish.
Consumer Satisfaction Questionnaire | 3 months
  Consumer satisfaction will be measured using an adapted version of a measure that has been used in other brief motivational interviewing interventions (Stormshak et al., 2005). Participants will reflect and report on their perceived quality of the modules they acccess and home practice. At the end of the program, participants will receive the adapted consumer satisfaction questionnaire to report their satisfaction.
Parenting Sense of Competency | baseline, 3 months, 6 months
  The Parenting Sense of Competency Scale (PSOC) will be used to measure parent efficacy. PSOC is a 19-item self-report measure that asks parents to what extent they agree or disagree with the statements regarding their parenting. PSOC has two subscales, including parent Self-efficacy (e.g., "Even though being a parent could be rewarding, I am frustrated while my child is at his/her present age.") and parent satisfaction (e.g., "I would make a good role model for new parents who needed to learn what it takes to be a good parent."). PSOC has overall good internal consistency (Cronbach's alpha = 0.82), and has been used with Spanish speaking parents. Parents respond on a 6-point Likert scale (1 = strongly agree to 6 = strongly disagree).
Latino Immigration Family Socialization Scale | baseline, 3 months, 6 months
  Socialization will be measured by the Latino Immigrant Family Socialization Scale (LIFS). LIFS is a 27-item self-report measure that contains six subscales, including adapt (5 items; e.g., "Encourage TC to learn to live with discrimination"), advocate (4 items; e.g., "Tell TC to seek help when he or she is discriminated"), cultural socialization (5 items; e.g., "Talk to TC about his or her roots and heritage"), educate about nativity and documentation (5 items; e.g., "Talk to TC about differences in rights based on immigration status"), value diversity (5 items; e.g., "Talk to TC about differences in cultures"), and promote mistrust (5 items; e.g., "Advice TC to be careful of people who are members of other racial or ethnic groups"). For each item, parents report how often they use these strategies on a 5-point Likert scale (1 = never to 5 = always). LIFS has been validated and shown acceptable internal consistencies (Cronbach's alphas > 0.70).
Adaptation of Parenting Young Children | baseline, 3 months, 6 months
  The Parenting Young Children Measure, which has been used with middle school children, will be used to measure support of good behavior (e.g., "Notice and praise your child's good behavior?"), setting limits (e.g., "Stick to your rules and not change your mind?"), and proactive parenting (e.g., "Give reasons for your requests?"). Each scale had 7 items, and parents self report using a Likert scale from 1 (not at all) to 7 (most of the time). These three scales have been validated, and these subscales have shown good internal consistency (Cronbach's alphas ranged from 0.79 to 0.85. This has been translated into Spanish in prior FCU studies.

SECONDARY OUTCOMES:
Strengths and Difficulties Questionnaire | baseline, 3 months, 6 months
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioral screening tool used to assess emotional and social well-being in children and adolescents. It evaluates five key areas-emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship issues, and prosocial behavior-providing a balanced view of both strengths and challenges. This measure will identify areas where the intervention has improved internalizing and externalizing behaviors.
CRAFFT | baseline, 3 months, 6 months
  The CRAFFT is well-used adolescent substance use screener for adolescents 12-21 for clinical use. Example items include, "Do you ever use drugs or alcohol while you are by yourself (alone)?" and "Have you ever gotten in trouble while you were using drugs and alcohol?" The CRAFFT has been shown to predict DSM-5 substance use disorders among adolescents. Chronbach's alpha was α = .79 and the screener has been validated in Spanish.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Doty, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
External researchers will have access to de-identified, individual-level data, and members of the general public will have access to metadata, descriptive data, and summary data. External researcher requests for individual-level data must be accompanied by a signed Data Use Agreement, and researchers must document that they are working under an institution with a Federal Wide Assurance (FWA). University of Oregon Information Services staff will develop and maintain the enclave to host and provide access to de-identified study data. The data enclave will be accessible to qualified researchers through a web portal that has capabilities to send and receive data by using encrypted secure transmission protocols.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual-level data will be released 12 months after the final participant has completed a given wave of data collection. This will allow time for data cleaning, and also provides a brief window for the investigative team to analyze and publish key findings prior to sharing the data, but still makes the data available to external researchers in a timely manner. After the grant award ends, if no additional external support is available to provide access to the data, the investigators will partner with the University of Oregon Libraries to host the data enclave and provide access to the data in perpetuity.
Access Criteria: External researcher requests for de-identified individual-level data must be accompanied by a signed Data Use Agreement, and researchers must document that they are working under an institution with a Federal Wide Assurance (FWA). If no additional external support is available to provide access to the data, we will partner with the University of Oregon Libraries to host the data enclave and provide access to the data.
URL: https://researchguides.uoregon.edu/data-management/dmp

REFERENCES:
- [Background] Mauricio AM, Hails KA, Caruthers AS, Connell AM, Stormshak EA. Family Check-Up Online: Effects of a Virtual Randomized Trial on Parent Stress, Parenting, and Child Outcomes in Early Adolescence. Prev Sci. 2024 Sep 24. doi: 10.1007/s11121-024-01725-3. Online ahead of print. PMID 39316242
- [Background] Stormshak EA, Seeley JR, Caruthers AS, Cardenas L, Moore KJ, Tyler MS, Fleming CM, Gau J, Danaher B. Evaluating the efficacy of the Family Check-Up Online: A school-based, eHealth model for the prevention of problem behavior during the middle school years. Dev Psychopathol. 2019 Dec;31(5):1873-1886. doi: 10.1017/S0954579419000907. PMID 31407644